CLINICAL TRIAL: NCT07215923
Title: A First in Human, Double-Blind, Placebo-Controlled, Randomized Evaluation of Single Ascending Doses of ATI-1013, a Human Monoclonal Antibody to Nicotine in Healthy Smokers
Brief Title: A First in Human Single Ascending Dose (SAD) Study of ATI-1013 in Healthy Smokers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Antidote Therapeutics, Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-1013-001; 5U01DA058547-03 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Thromboangiitis Obliterans (Buerger's Disease)
Keywords: ATI-1013; Anti-nicotine monoclonal antibody; Nicotine dependence; Tobacco use disorder; Smoking cessation; Smoking reduction; Vascular disease; Phase 1; Healthy adult smokers
MeSH Terms: conditions — Thromboangiitis Obliterans; Tobacco Use Disorder; Smoking Cessation; Smoking Reduction; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATI-1013 (0.2 g) (Experimental): Single-ascending-dose Cohort 1. Participants receive a single intravenous (IV) infusion of ATI-1013 0.2 g on Day 1. Randomization within the cohort is 4:1 (ATI-1013:placebo).
  Interventions: Biological: ATI-1013 (0.2 g); Other: Placebo
- ATI-1013 (0.8 g) (Experimental): Single-ascending-dose Cohort 2. Participants receive a single IV infusion of ATI-1013 0.8 g on Day 1. Randomization 4:1 (ATI-1013:placebo).
  Interventions: Biological: ATI-1013 (0.8 g); Other: Placebo
- ATI-1013 (3.2 g) (Experimental): Single-ascending-dose Cohort 3. Participants receive a single IV infusion of ATI-1013 3.2 g on Day 1. Randomization 4:1 (ATI-1013:placebo).
  Interventions: Biological: ATI-1013 (3.2 g); Other: Placebo

INTERVENTIONS:
Biological: ATI-1013 (0.2 g) — Single intravenous (IV) infusion of ATI-1013, 0.2 g total dose.
  Arms: ATI-1013 (0.2 g)
Biological: ATI-1013 (0.8 g) — Single IV infusion of ATI-1013, 0.8 g total dose.
  Arms: ATI-1013 (0.8 g)
Biological: ATI-1013 (3.2 g) — Single IV infusion of ATI-1013, 3.2 g total dose.
  Arms: ATI-1013 (3.2 g)
Other: Placebo — Matching placebo (vehicle) IV infusion.

SUMMARY:
This study is a first-in-human clinical trial of drug ATI-1013, in healthy adult cigarette smokers. The main questions it aims to answer are to learn about the safety of drug ATI-1013, how long drug ATI-1013 remains within the body, does drug ATI-1013 trigger an immune response, and the effects of drug ATI-1013 on nicotine levels within the body.

The clinical trial will compare drug ATI-1013 to a placebo (a look-alike substance that contains no drug) to see if drug ATI-1013 has comparable safety.

Participants will have a Screening visit (Day -28 to -3) and will be admitted on Day -2. Each participant will receive one intravenous (IV) infusion of ATI-1013 or placebo (Day 1). Participants will remain in-clinic for at least 48 hours post-dose and return for follow-up visits on Days 7, 21, 42, 56, and 84, with telephone check-ins on Days 5, 14, 28, and 70. Participants will keep a diary of their cigarette use and smoking behaviors.

ELIGIBILITY:
Inclusion Criteria

1. Provides written informed consent before any study procedures
2. Age 23 to 59 years, inclusive
3. Body weight ≥50 kg at Screening
4. Body mass index (BMI) 18.5-29.9 kg/m² at Screening
5. In good health with no medically significant conditions, in the opinion of the Investigator
6. Current smoker, ≥10 cigarettes per day for ≥2 years, with no abstinence >6 months
7. Female participants must agree not to donate ova during the study and for 90 days after dosing
8. Female participants of childbearing potential must use an acceptable, effective method of birth control from 30 days prior to Screening through 90 days after dosing
9. Female participants of non-childbearing potential must be surgically sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation) or postmenopausal (≥1 year without menses)
10. Male participants must agree to use contraception and not donate sperm for 90 days after dosing
11. Willing to abstain from all other tobacco products from Day -2 through Day 84
12. Willing to abstain from all other nicotine products from Day -2 through Day 84
13. Willing to abstain from smoking regular cigarettes:

    1. Approximately 18 hours from evening of Day -2
    2. Approximately 42 hours from evening of Day -1

Exclusion Criteria

1. Pregnant, breastfeeding, or planning pregnancy
2. Positive serum pregnancy test at Screening or urine pregnancy test on Day -2 (women only)
3. Prior exposure to any anti-nicotine vaccine or antibody
4. Use of mentholated tobacco products within 30 days before Screening, unwilling to refrain during the study
5. History of severe allergic reaction to antibodies or vaccines (including Guillain-Barré syndrome)
6. Received any vaccination within 90 days prior to Screening
7. Clinically significant allergic adverse reaction (seasonal allergies allowed)
8. Use of systemic steroids or immunomodulating drugs within 90 days (inhaled steroids allowed)
9. History of cancer (except treated basal/squamous cell skin cancer), HIV, other immunodeficiency, or autoimmune disease
10. History of drug (excluding nicotine) or alcohol use disorder (DSM-5 criteria)
11. Clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, or psychiatric disorder, as determined by the Investigator
12. Clinically significant abnormal clinical chemistry, hematology, or urinalysis at Screening or Day -2, in the opinion of the Investigator
13. COVID-19 within the past 6 months or ongoing symptoms likely attributable to COVID-19
14. Use of varenicline, bupropion, nicotine replacement therapy (NRT), or other anti-smoking pharmacologic treatments (including off-label nortriptyline, clonidine, or cytisinicline) within 90 days prior to Screening
15. Received an investigational product within 30 days (90 days for biologics) or 5 half-lives (whichever is longer) prior to Screening
16. Exhaled carbon monoxide (CO) <8 ppm at Screening
17. Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody at Screening
18. Positive urine alcohol test at Screening and/or Day -2
19. Positive urine drug test (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids) at Screening and/or Day -2
20. Unwilling to abstain from xanthine-containing products (coffee, tea, cola, chocolate, energy drinks) within 24 hours prior to admission until discharge
21. Unwilling to abstain from alcohol or alcohol-containing products within 24 hours prior to admission until discharge
22. Significant blood donation or blood loss >500 mL within 56 days before Screening
23. Plasma donation or loss within 30 days prior to Screening through Day 84
24. Hypersensitivity to the study drug, its excipients, or similar products
25. Unable or unwilling to comply with protocol requirements, restrictions, or instructions
26. Currently enrolled in another clinical study

Ages: 23 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of all adverse events (AEs) | Day 1 through Day 84
  Incidence of all adverse events (AEs), including infusion-related reactions (IRRs) and injection site reactions.
Development of Anti-Drug Antibodies | Baseline (Day -1) through Day 84
  Presence of anti-ATI-1013 antibodies following a single intravenous infusion.

SECONDARY OUTCOMES:
Pharmacokinetics of ATI-1013 Maximum Concentration (Cmax) | Day 1 through Day 84
  Serum ATI-1013 maximum concentration.
Pharmacokinetics of ATI-1013 Time to Maximum Concentration (Tmax) | Day 1 through Day 84
  Serum ATI-1013 time to maximum concentration.
Pharmacokinetics of ATI-1013 Area Under the Curve (AUC) | Day 1 through Day 84
  Serum ATI-1013 area under the curve.
Pharmacokinetics of ATI-1013 Half-life (t1/2) | Day 1 through Day 84
  Serum ATI-1013 half-life.
Physiologic Responses to Nicotine (Skin Temperature) | Day -1 and Day 2
  Changes in physiologic responses to nicotine, including skin temperature (°F).
Physiologic Responses to Nicotine (Heart Rate) | Day -1 and Day 2
  Changes in physiologic responses to nicotine, including heart rate (beats per minute).
Physiologic Responses to Nicotine (Plasma Epinephrine) | Day -1 and Day 2
  Changes in physiologic responses to nicotine, including plasma epinephrine (picograms per milliliter (pg/mL)).
Physiologic Responses to Nicotine (Blood Pressure) | Day -1 and Day 2
  Changes in physiologic responses to nicotine, including blood pressure (mmHg).
Withdrawal Symptoms Minnesota Tobacco Withdrawal Scale (MTWS) | Day -1 and Day 2
  Self-reported withdrawal symptoms measured using the MTWS. (Minimum Value 0; Maximum Value 68; Higher score is a stronger withdrawal effect)
Subjective/Psychological Effects of Nicotine Drug Effect Questionnaire (DEQ) | Day -1 and Day 2
  Self-reported subjective/psychological effects of nicotine using the DEQ (visual analogue scale from not at all to extremely, measure in millimeters; Higher score is a stronger effect of the cigarette).
Subjective/Psychological Effects of Nicotine Modified Cigarette Evaluation Questionnaire (mCEQ) | Day -1 and Day 2
  Self-reported subjective/psychological effects of nicotine using the mCEQ (Minimum Value 12; Maximum Value 84; Higher score is a stronger addiction).
Total Nicotine Levels | Baseline through Day 84
  Blood concentrations of total nicotine.
Free Nicotine Levels | Baseline through Day 84
  Blood concentrations of free nicotine.
ATI-1013-Bound Nicotine Levels | Baseline through Day 84
  Blood concentrations of ATI-1013-bound nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kalnik, PhD, Study Chair — Antidote Therapeutics, Inc
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No